CLINICAL TRIAL: NCT00005850
Title: Fluoxetine in Stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC): A Phase II Pilot Study to Improve Quality of Life During Chemotherapy
Brief Title: Combination Chemotherapy Plus Fluoxetine in Treating Patients With Advanced or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-119802; U10CA031946 (NIH); CLB-119802; CDR0000067871 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Anxiety Disorder; Depression; Fatigue; Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; fatigue; anxiety disorder; depression
MeSH Terms: conditions — Anxiety Disorders; Depression; Fatigue; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cisplatin; Fluoxetine; Gemcitabine

ARMS (1):
- gemcitabine + cisplatin + fluoxetine (Experimental): Patients receive gemcitabine and cisplatin. Treatment repeats every 21 days for a total of six cycles. Patients receive fluoxetine for 7 weeks. Further use of fluoxetine is at the discretion of the patient and physician.
  Interventions: Drug: cisplatin; Drug: fluoxetine; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: cisplatin — 80 mg/m2 administered by intravenous (IV) over 30 minutes on Day 1 following the gemcitabine infusion. Treatment repeated every 21 days for a total of 6 cycles.
Drug: fluoxetine — 10 mg PO QD (by mouth once daily) starting on week 2 (day 8) and continuing for 7 weeks (days 8-57). After 7 weeks of fluoxetine treatment (day 57), further use of fluoxetine is at the discretion of the patient and physician.
Drug: gemcitabine hydrochloride — 1000 mg/m2 intravenous (IV) administered by IV over 30 minutes on days 1 and 8. Repeat treatment every 21 days for a total of 6 cycles.

SUMMARY:
This trial is designed to test the efficacy of fluoxetine to improve patient's quality of life during chemotherapy. An innovative application of a selective serotonin reuptake inhibitor may modulate the effects of fatigue, anxiety and depression which worsen quality of life.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objectives:

1. To preliminarily test the efficacy of fluoxetine to improve the quality of life of patients with advanced non-small cell lung cancer receiving chemotherapy by decreasing anxiety, depression and fatigue.
2. To test the feasibility of conducting a multi-center clinical trial of fluoxetine administered by oncologists concurrently with chemotherapy in patients with non-small cell lung cancer.

Secondary Objectives:

1. To describe the tumor response rate associated with the administration of gemcitabine/cisplatin in patients with advanced non-small cell lung cancer.
2. To describe the overall survival and failure-free survival associated with the administration of gemcitabine/cisplatin.
3. To describe the toxicity associated with the administration of gemcitabine/cisplatin.

ELIGIBILITY:
Eligibility Criteria:

1. Histologic Documentation: All patients must have histologically or cytologically documented, non-small cell carcinoma of the lung (adenocarcinoma, large cell, squamous, or mixtures of these types).
2. Extent of Disease: Stage IIIB/IV cancer by the international staging system or any Stage I-IIIA otherwise eligible patient with recurrent or progressive NSCLC after surgery or radiotherapy.

   * Patients with Stage IIIB because of a malignant pleural effusion, supraclavicular node involvement, or contralateral hilar nodes are eligible (IIIB patients eligible for CALGB protocols of combined chemotherapy and chest irradiation are not eligible.
   * Patients with known CNS metastases are not eligible.
3. Measurable or Non-Measurable Disease

   * Measurable Disease: Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan.
   * Non-measurable Disease: Only those non-measurable disease patients with ill-defined masses associated with post-obstructive changes and diffuse parenchymal malignant disease are eligible. All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions, are not eligible.

   Lesions that are considered non-measurable include the following:
   * Bone lesions
   * Leptomeningeal disease
   * Ascites
   * Pleural/pericardial effusion
   * Abdominal masses that are not confirmed and followed by imaging techniques
   * Cystic lesions
4. Prior Treatment:

   * No prior chemotherapy.
   * ≥ 2 weeks since radiation therapy.
   * No antidepressant treatment (eg, selective serotonin reuptake inhibitors, tricyclics, novel antidepressants, St. John's Wort or monoamine oxidase inhibitors) currently or within the last month.
5. If the patient requires pain medication, pain must be managed with non-codeine preparations, including but not limited to: acetaminophen, any morphine based preparation (short or long acting), hydromorphone, fentanyl, levorphanol or methadone.
6. CTC Performance Status 0-1.
7. Non-pregnant and non-nursing because of significant risk to the fetus/infant.
8. Required Initial Laboratory Data:

   * Granulocytes ≥ 1,500/µl
   * Platelet count ≥ 100,000/µl
   * Serum creatinine ≤ 1.5 mg/dl or Calculated CrCl ≥ 60 ml/min
   * Bilirubin ≤ 2.0 x Upper Limit of Normal (ULN)
   * Serum glutamic oxaloacetic transaminase (SGOT) ≤ 2.0 x ULN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Change in the MHI-17 global psychological distress subscale | Up to 8 weeks
Overall survival | Up to 2 years post-treatment
Failure-free survival | Up to 2 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Donna Greenberg, MD, Study Chair — Massachusetts General Hospital
Locations (43):
- United States (42):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Medical Center, Boston, Massachusetts
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan, Puerto Rico